CLINICAL TRIAL: NCT03636321
Title: Randomized Controlled Clinical Trial Of Stented Versus Stentless Biliary Anastomosis In Living Donor Liver Transplantation
Brief Title: Stented Biliary Anastomosis in Living Donor Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Mstafa Hassan Sewefy (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Alaa Mstafa Hassan Sewefy, professor, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS.fac.med.55
Record Dates: First submitted 2018-08-02; First posted 2018-08-17 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Liver Transplant
Keywords: living donor liver transplantation; intraductal stent; biliary complications after liver transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intraductal stent (Experimental): in this group ,patients candidate for living donor liver transplantation duct to duct biliary anastomosis with internal biliary stent
  Interventions: Procedure: living donor liver transplantation with internal biliary stent
- stentless (Active Comparator): in this group ,patients candidate for living donor liver transplantation duct to duct biliary anastomosis will done without internal biliary
  Interventions: Procedure: living donor liver transplantation with internal biliary stent

INTERVENTIONS:
Procedure: living donor liver transplantation with internal biliary stent — living donor liver transplantation without internal biliary stent

SUMMARY:
Determination of biliary complications in stented group compared to duct to duct anastomosis without stent

DETAILED DESCRIPTION:
30 patients included in the study. patients will be randomly allocated in two equal groups. In group A anastomosis will be done on intraductal stent and in group B anastomosis done without stent .the patients will be followed for one year to compare the result of two groups as regard biliary complications.

ELIGIBILITY:
Inclusion Criteria:

* adult patients eligible for a liver transplantation
* patients' written informed consent signed.

Exclusion Criteria:

* biliary reconstruction requires a hepatico-jejunostomy for anatomical/biliary disease reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
biliary complications after living donor liver transplantation | one year
  incidence of biliary complications after living donor liver transplantation

SECONDARY OUTCOMES:
biliary complications | one year
  types of biliary complications
biliary related mortality | one year
  mortality
rate of cholangitis | 3 months
  rate of cholangitis
hospital stay | one month
  hospital stay
time 2 biliary complications | one year
  time 2 biliary complications

OTHER OUTCOMES:
skeletonization of duct | 10 hours
  skeletonization of duct

CONTACTS AND LOCATIONS:
Locations (1):
- Air force spcialized hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided